CLINICAL TRIAL: NCT05703490
Title: An Innovative Platform for Objective Monitoring of Instrumental Activities of Daily Living
Status: Terminated | Type: Observational
Why Stopped: The PI has moved to another institution
Sponsor: Bijan Najafi, PhD (Other)
Collaborators: BioSensics (Industry)
Responsible Party: Sponsor-Investigator, Bijan Najafi, PhD, Professor of Surgery, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Other Study IDs: H-43413
Record Dates: First submitted 2022-10-11; First posted 2023-01-30 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Dementia; Cognitive Impairment; Alzheimer Disease
Keywords: dementia; activities of daily living; MCI; Telehealth; Smart home; IOT
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cognitive Impaired Group: older adults (age 50 years and older) with either clinical diagnosis of cognitive impairment or determined to have cognitive impairment based on Montreal Cognitive Assessment (MoCA) Test, score of 26 or lower
  Interventions: Diagnostic Test: IADLSys system
- Cognitive Intact Group: Older adults age matched with Cognitive Impaired Group with MoCA score of greater than 26
  Interventions: Diagnostic Test: IADLSys system

INTERVENTIONS:
Diagnostic Test: IADLSys system — Subjects will receive IADLSys system which includes interactive tablet and 5 paired pTAGs (bluetooth sensors to attach to objects of interest at home). The pTAGs monitor activities of daily living to assess if they are being completed and communicate with the tablet to keep record of interactions. We anticipate IADLSys enables to distinguish between groups with and without cognitive impairment and determine the severity of cognitive impairment in the cognitive impaired group.

SUMMARY:
Difficulties in performing instrumental activity of daily living (IADL) is often an indicator of cognitive decline in older adults, and monitoring IADL and daily functioning can assist in early diagnosis of dementia. The current methods for assessment of IADL are often restricted to a single domain assessment (e.g. managing medication), or rely on subjective reporting by the patient or caregivers. Patients with mild AD typically lack awareness of their IADL deficits and generally overestimate their functional capacity. Proxies are also not always a reliable source of information, as they have a tendency to over or underestimate IADL deficits. In some cases, a proxy is not available or does not have enough knowledge about the patient's functional capacity. Direct measures taken during performance of IADL-related tasks in the clinic have better validity and do not suffer from reporter bias. However, they allow observation of only a small set of tasks and, even then, are quite time-consuming. To date, there are no objective methods for continuous and remote monitoring and assessment of IADL. The National Institute on Aging (NIA) has identified this need and released a specific request for SBIR/STTR applications. In response, BioSensics, in collaboration with Baylor College of Medicine (BCM), proposes to develop and commercialize a robust system for objective and continuous remote monitoring of IADL. This innovative platform, called IADLSys, will detect the timing and type of IADL for a wide range of daily functions, and will also monitor the user's physical activity and life-space.

DETAILED DESCRIPTION:
This innovative platform, called IADLSys, will detect the timing and type of IADL for a wide range of daily functions, and will also monitor the user's physical activity and life-space. There are two key aspects of the technology: 1) physical tags (pTAGs): a series of sensors that can be attached to various objects to monitor the user's interaction with these objects, 2) PAMSys+: a pendant wearable sensor to monitor physical activity and the user's proximity to the pTAGs. As a part of this development, the investigators will create a base station to collect and transfer data from wireless sensors and wearable pendant to a secure backend cloud. A secure website will be developed to allow caregivers and medical professionals access and view collected data. For the validation of the platform, the investigators will recruit a total of 100 participants with and without cognitive impairment (50 subjects per group). Eligible subjects will undergo one week observational study while using the system at home. The investigators hypothesize that monitoring performance of IADLs, their timing, as well as other metrics like life space size and patterns of physical activity can discriminate between groups. Furthermore, the acceptability, perception of benefit, and ease of use of IADLSys will be assessed using a technology acceptance model questionnaire (TAM) adopted for tele-health applications

ELIGIBILITY:
Inclusion Criteria:

* 50 years or older
* Ambulatory and are living independently in a residential home with a caregiver/informant
* Willing and able to provide informed consent

Exclusion Criteria:

* Under 50 years
* immobility or inability to engage in IADL that are essential for independent living
* Patients with any clinically significant medical or psychiatric condition
* Recent stroke over last 6 months
* major hearing/visual impairment
* any acute diagnosis that may impact IADL (e.g., fracture, foot ulcer, recent surgery, etc)
* residing in a nursing home or are receiving hospice care
* inability to communicate in English
* are unlikely to fully comply with the follow-up protocol

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ambulatory older adults (over 50 years old) with and without cognitive impairment.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Medication adherence | 1 week
  Medication adherence is assessed by self-report as well as IADLSys
Cognitive function | Baseline
  Cognitive function is assessed by Montreal Cognitive Assessment (MoCA) Test. A score of 26 or lower is considered as cognitive impaired.

SECONDARY OUTCOMES:
Changes in acceptability, perception of benefit, and ease of use of IADLSys System from baseline to follow up | baseline, 1 week
  Acceptability, perception of benefit, and ease of use will be assessed using Technology Acceptance Model questionnaire (TAM) adopted for tele-health applications. Initial opinions and scores from baseline will be compared to the answers at 1 week follow up.
History of fall | Baseline
  Self report history of falls will be documented at baseline
Depression | Baseline
  Depression is assessed by Center for Epidemiologic Studies Depression Scale (CES-D). Score ranges from 0 to 60, higher the score indicates presence of depression.
Life Space | one week
  The Life Space Questionnaire is a measure of the extent of mobility of older adults. Score ranges from 0-9, with higher score indicating the particpant uses more of their space regularly.
Adherence to physical activity monitoring from baseline to follow up | 1 week
  Adherence to physical activity monitoring by wearing a validated pendant sensor from baseline to 1 week will be assessed. Physical activity will be quantified by measuring number of taken steps per day and will be measured using a validated wearable sensor named PAMSys. Monitoring of physical activity will be done for 1 week from baseline to 1 week follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee M, Mishra RK, Momin A, El-Refaei N, Bagheri AB, York MK, Kunik ME, Derhammer M, Fatehi B, Lim J, Cole R, Barchard G, Vaziri A, Najafi B. Smart-Home Concept for Remote Monitoring of Instrumental Activities of Daily Living (IADL) in Older Adults with Cognitive Impairment: A Proof of Concept and Feasibility Study. Sensors (Basel). 2022 Sep 7;22(18):6745. doi: 10.3390/s22186745. PMID 36146095